CLINICAL TRIAL: NCT03510611
Title: A Pharmacokinetic Study in Chinese Healthy Male and Female Volunteers to Investigate the Effect of Food on the Pharmacokinetics of Ensartinib Capsules.
Brief Title: A Study to Investigate the Food Effect on the Pharmacokinetics of Ensartinib Capsules in Chinese Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BTP-44313
Record Dates: First submitted 2018-03-28; First posted 2018-04-27 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ensartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Period 1: fed control → Period 2: fasted control (Experimental): Period 1: administration of Ensartinib 225mg at 7:30am, 30 minutes after the breakfast；Period 2: administration of Ensartinib 225mg at 7:30am, without the breakfast
  Interventions: Drug: Ensartinib with fed or fasting
- Period 1: fasted control → Period 2: fed control (Experimental): Period 1: administration of Ensartinib 225mg at 7:30am, without the breakfast；Period 2: administration of Ensartinib 225mg at 7:30am, 30 minutes after the breakfast
  Interventions: Drug: Ensartinib with fed or fasting

INTERVENTIONS:
Drug: Ensartinib with fed or fasting — The two groups of subjects were given an equal dose of Ensartinib capsules (225 mg) after a single cross-over fasting or high-fat high-calorie diet in two different test cycles to examine the effect of food on the pharmacokinetics of Ensartinib.

SUMMARY:
The main objective of this study is to evaluate the Effect of Food on the Pharmacokinetics of Ensartinib Capsules.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the Effect of Food on the Pharmacokinetics of Ensartinib Capsules in Chinese Healthy Volunteers. In addition, the safety of Ensartinib Capsules in Chinese Healthy Volunteers who with High-fat meal or fasting state will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* age: 20 - 45 years;
* sex: male and female;
* body weight: Male ≥ 50 kg,female ≥ 45 kg, body mass index BMI (weight (kg)/height 2 (m2)) between 19-26 kg/m2 (including border);
* Healthy as judged by the investigator/subinvestigator based on the results of physical examinations and all lab tests;
* written informed consent;

Exclusion Criteria:

* Received any investigational drugs within 14 days before the screening test;
* Donated 200 mL of whole blood within 30 days before the screening test,or Donated 200 mL of whole blood during the study or within 30 days after completion of the study;
* Females who are lactating, pregnant, potentially child-bearing, or willing to get pregnant during the study period;
* History of drug or food allergies;
* Abnormal blood pressure or pulse，Abnormal laboratory tests;
* Participated in other clinical trials within 3 months before screening;
* Smoking and drinking within 3 months before screening or test results of smoke, alcohol, and drug abuse are positive;Positive for HBsAg, Hepatitis C virus (HCV) antibody, HIV antibody or syphilis antibody;Clinically apparent disease/infection within 1 month before screening;
* Positive for HBsAg, Hepatitis C virus (HCV) antibody, HIV antibody or syphilis antibody;
* Clinically apparent disease/infection within 1 month before screening;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) of Ensartinib | pre-dose(30minute),30min,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12,24,36,48,72,96,120hour
  The effect of food on Cmax after high fat diet and fasting Blood sampling over a 120 hour period post dose in all dosing sessions
Area under the plasma concentration versus time curve (AUC) of Ensartinib | pre-dose(30minute),30min,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12,24,36,48,72,96,120hour
  The effect of food on AUC after high fat diet and fasting Blood sampling over a 120 hour period post dose in all dosing sessions
Time of maximum concentration（Tmax）of Ensartinib | pre-dose(30minute),30min,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12,24,36,48,72,96,120hour
  The effect of food on Tmax after high fat diet and fasting Blood sampling over a 120 hour period post dose in all dosing sessions
Half life（T1/2）of Ensartinib | pre-dose(30minute),30min,1,1.5,2,2.5,3,3.5,4,4.5,5,6,8,12,24,36,48,72,96,120hour
  The effect of food on T1/2 after high fat diet and fasting Blood sampling over a 120 hour period post dose in all dosing sessions

SECONDARY OUTCOMES:
Percentage of adverse events | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 months
  Percentage of adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: zourong ruan, Study Chair — the Second Affiliated Hospital of Zhejiang University Medical College
Locations (1):
- The 1st Phase Clinical Research Center of the Second Affiliated Hospital of Zhejiang University Medical College, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No